CLINICAL TRIAL: NCT01188551
Title: Pain Management Following Myringotomy and Tube Placement: Intranasal Dexmedetomidine Versus Fentanyl
Brief Title: Dexmedetomidine Versus Fentanyl Following Pressure Equalization Tube Placement
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Joseph D. Tobias, Chairman Dept. of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB10-00377
Record Dates: First submitted 2010-08-24; First posted 2010-08-25 (Estimated); Results first posted 2014-04-01 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2014-02

CONDITIONS: Chronic Otitis Media
Keywords: myringotomy; pressure equalization tubes
MeSH Terms: interventions — Dexmedetomidine; Fentanyl; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- dexmedetomidine w/ midazolam (Experimental): Midazolam 0.5 mg/kg given orally pre-op and 1 dose of dexmedetomidine 1mcg/kg given intranasally in OR.
  Interventions: Drug: Dexmedetomidine; Drug: Midazolam
- fentanyl w/ midazolam (Active Comparator): Midazolam 0.5 mg/kg given orally pre-op and 1 dose of fentanyl 2mcg/kg given intranasally in OR.
  Interventions: Drug: Fentanyl; Drug: Midazolam
- dexmedetomidine w/o midazolam (Experimental): 1 dose of dexmedetomidine 1mcg/kg given intranasally in OR without any pre-medication.
  Interventions: Drug: Dexmedetomidine
- fentanyl w/o midazolam (Active Comparator): 1 dose of fentanyl 2mcg/kg given intranasally in the OR without any pre-medication.
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Dexmedetomidine — dexmedetomidine (1 µg/kg) will be administered intranasally
  Other Names: Precedex
  Arms: dexmedetomidine w/ midazolam; dexmedetomidine w/o midazolam
Drug: Fentanyl — fentanyl (2 µg/kg) will be administered intranasally
  Arms: fentanyl w/ midazolam; fentanyl w/o midazolam
Drug: Midazolam — Sedative given pre-op.
  Other Names: Versed
  Arms: dexmedetomidine w/ midazolam; fentanyl w/ midazolam

SUMMARY:
This is a study to compare intranasal dexmedetomidine to intranasal fentanyl following anesthesia induction in patients undergoing myringotomy and placement of pressure equalization (PE) tubes in providing analgesia and smoothing emergence from general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* functional status as assigned by the American Society of Anesthesiology (ASA) classification of I or II (no or minimal co-morbid disease)
* patients scheduled for placement of bilateral myringotomy tubes

Exclusion Criteria:

* history of allergy to either dexmedetomidine or fentanyl
* concomitant use of medications which may exaggerate the HR response of dexmedetomidine including digoxin or β-adrenergic antagonists.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Background] Tobias JD. Dexmedetomidine: applications in pediatric critical care and pediatric anesthesiology. Pediatr Crit Care Med. 2007 Mar;8(2):115-31. doi: 10.1097/01.PCC.0000257100.31779.41. PMID 17273114
- [Background] Yuen VM, Irwin MG, Hui TW, Yuen MK, Lee LH. A double-blind, crossover assessment of the sedative and analgesic effects of intranasal dexmedetomidine. Anesth Analg. 2007 Aug;105(2):374-80. doi: 10.1213/01.ane.0000269488.06546.7c. PMID 17646493

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the outpatient ENT surgery service at Nationwide Children's Hospital.
Groups:
- Dexmedetomidine w/ Midazolam: Midazolam given orally pre-op and dexmedetomidine given intranasally in OR.
- Fentanyl w/ Midazolam: Midazolam given orally pre-op and fentanyl given intranasally in OR.
- Dexmedetomidine w/o Midazolam: Dexmedetomidine given intranasally in OR without any pre-medication.
- Fentanyl w/o Midazolam: Fentanyl given intranasally in the OR without any pre-medication.
Period: Overall Study
Arm/Group | Dexmedetomidine w/ Midazolam | Fentanyl w/ Midazolam | Dexmedetomidine w/o Midazolam | Fentanyl w/o Midazolam
Started | 25 | 25 | 25 | 25
Completed | 24 | 25 | 25 | 25
Not Completed | 1 | 0 | 0 | 0
Not completed — Pharmacy issues | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine w/ Midazolam | Fentanyl w/ Midazolam | Dexmedetomidine w/o Midazolam | Fentanyl w/o Midazolam | Total
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 25 | 25 | 25 | 25 | 100
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.14 (1.01) | 3 (2.02) | 2.98 (1.87) | 2.22 (1.16) | 3 (1.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 9 | 5 | 38
  Male | 15 | 11 | 16 | 20 | 62
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 25 | 25 | 100

OUTCOME MEASURES:

1. Primary Outcome: FLACC Behavioral Pain Assessment Scale Scores
Description: FLACC Behavioral Pain Assessment Scale: each of the five categories (F) Face, (L) Legs, (A) Activity, (C) Cry, (C) Consolability is scored from 0-2, which results in a total score between 0 and 10.
  0 = Relaxed and comfortable 1-3 = Mild discomfort 4-6 = Moderate pain 7-10 = Severe discomfort or pain or both
Time Frame: 30 mins. post-op
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dexmedetomidine w/ Midazolam | Fentanyl w/ Midazolam | Dexmedetomidine w/o Midazolam | Fentanyl w/o Midazolam
Number analyzed (Participants) | 24 | 25 | 25 | 25
units on a scale | 5 (4.19) | 3 (3.60) | 1 (2.20) | 2 (2.92)

2. Secondary Outcome: Recovery From General Anesthesia
Description: Post-anesthesia recovery score: Aldrete The Aldrete scoring system takes into account the patient's ability to move, respiration, circulation, consciousness, and oxygen saturation. A maximum of two points are awarded in each category and a score of 9 or 10 is required for discharge.
Time Frame: 30 mins. post-op
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dexmedetomidine w/ Midazolam | Fentanyl w/ Midazolam | Dexmedetomidine w/o Midazolam | Fentanyl w/o Midazolam
Number analyzed (Participants) | 24 | 25 | 25 | 25
units on a scale | 8.67 (1.33) | 9 (0.96) | 9.25 (0.94) | 9.5 (0.74)

ADVERSE EVENTS:
Arm/Group | Dexmedetomidine w/ Midazolam | Fentanyl w/ Midazolam | Dexmedetomidine w/o Midazolam | Fentanyl w/o Midazolam
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes